CLINICAL TRIAL: NCT01334008
Title: Development and Validation of a Circulating Tumor DNA Detection Technique in Patients With Metastatic Choroidal Melanoma
Brief Title: Study of Circulating Tumoral DNA in Metastatic Choroidal Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2010-02
Record Dates: First submitted 2011-03-31; First posted 2011-04-12 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Choroidal Melanoma, Diffuse
Keywords: Circulating tumor DNA; Choroidal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood sampling (Other)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — 30ml of patient peripherical blood will be collected

SUMMARY:
Circulating tumor DNA detection and quantification in patients with metastatic choroidal melanoma.

DETAILED DESCRIPTION:
Technique development: In first step, the different available techniques will be evaluated for specificity and sensibility using serial dilutions of cell lines with or without GNAQ mutation.

Validation: The tumor DNA detection rate will be estimated from metastatic uveal patient's blood. The investigators will study 40 patients to obtain at least 15 patients bearing a GNAQ mutation in the primitive tumor or in metastasis. With those 15 patients, the investigators will determinate the most sensitive technique and the best cost/efficiency ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years.
* Patient with a metastatic choroidal melanoma.
* Patient with tumor or metastasis available for GNAQ (Guanine nucleotide blinding protein) status characterization.
* Patient able to stand a blood collection.
* Signed written informed consent approved by competent authority and ethic committee.

Exclusion Criteria:

* Patient without social protection/insurance.
* Current pregnancy and lactation.
* All social, medical, psychological, situations making the study impossible.
* Person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Assessment and development of circulating tumor DNA detection techniques | 2 years
  Quantification of circulating tumor DNA in blood samples. Results expressed in number of samples where circulating DNA is present.

SECONDARY OUTCOMES:
Detection technique comparison (PAP (pyrophosphorolysis activated polymerisation), BEAMing, NGS(next sequencing generation)) in terms of feasibility, robustness, sensitivity and cost. | 2 years
  The methods of detection which will be used such as the BEAMing, the PAP (Pyrophosphorolysis-activated polymerization) and NGS (next sequencing generation)is techniques of a big specificity capable of detecting a mutant copy among 1.104 wild copies for the BEAMing, 2.109 for the PAP and 1.105 for the NGS. The sensibility of these techniques is limited by the quantity of genomic DNA which we can extract from the sample of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PIPERNO-NEUMANN, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Bidard FC, Madic J, Mariani P, Piperno-Neumann S, Rampanou A, Servois V, Cassoux N, Desjardins L, Milder M, Vaucher I, Pierga JY, Lebofsky R, Stern MH, Lantz O. Detection rate and prognostic value of circulating tumor cells and circulating tumor DNA in metastatic uveal melanoma. Int J Cancer. 2014 Mar 1;134(5):1207-13. doi: 10.1002/ijc.28436. Epub 2013 Sep 3. PMID 23934701